CLINICAL TRIAL: NCT02604147
Title: Inspiratory Muscle Training in Wheelchair Basketball Players: Effects on Physical Performance and Cardiopulmonary Variables
Brief Title: Inspiratory Muscle Training in Wheelchair Basketball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Metodista de Piracicaba (Other)
Responsible Party: Principal Investigator, Raphael do Nascimento Pereira, MsC., Universidade Metodista de Piracicaba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UNIMEP
Record Dates: First submitted 2015-09-25; First posted 2015-11-13 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Respiratory Muscles; Breathing Exercises; Athletic Performance; Athletes; Aerobic Capacity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Simulated inspiratory muscle training (Sham Comparator): Inspiratory muscle training with load of 15% of maximal inspiratory pressure.
  Interventions: Device: Inspiratory pressure-threshold muscle training device.
- Inspiratory muscle training group (Experimental): Inspiratory muscle training with initial load of 50% of maximal inspiratory pressure.
  Interventions: Device: nspiratory pressure-threshold muscle training device.

INTERVENTIONS:
Device: Inspiratory pressure-threshold muscle training device. — The participants who will be allocated in this simulated intervention group will have to do a simulated inspiratory muscle training protocol through the inspiratory muscle exerciser POWERbreathe, model Sports Plus Heavy Resistance (POWERbreathe; HAB International Ltd., Warwickshire, United Kingdom) for 12 weeks five times at week and twice daily, with a load of 15% of maximal inspiratory pressure without progression. In each session will be requested to the volunteers make 30 slow breaths, which will be constantly supervised by the researchers.
  Other Names: POWERbreathe - model Sports Plus Heavy Resistance (HAB International Ltd., Warwickshire, United Kingdom).
  Arms: Simulated inspiratory muscle training
Device: nspiratory pressure-threshold muscle training device. — The participants who will be allocated in this intervention group will have to make a inspiratory muscle training protocol with progressive loads through the inspiratory muscle exerciser POWERbreathe, model Sports Plus Heavy Resistance (POWERbreathe; HAB International Ltd., Warwickshire, United Kingdom) for 12 weeks five times at week and twice daily, with an initial load of 50% of maximal inspiratory pressure, progressing to 60% after the fourth week, and 70% after the octave week. In each session will be requested to volunteers who performed 30 maximal and prolonged inspiration, maintaining the diaphragmatic breathing, which will be constantly supervised by the researchers.
  Other Names: POWERbreathe - model Sports Plus Heavy Resistance (HAB International Ltd., Warwickshire, United Kingdom).
  Arms: Inspiratory muscle training group

SUMMARY:
Investigate the effects of Inspiratory Muscle Training on the physical performance and cardiorespiratory variables of wheelchair basketball players.

DETAILED DESCRIPTION:
The respiratory system has been touted as a limiting factor of physical performance during high intense physical exercises. This limitation is related, among other things, with the fatigue of respiratory muscles. The fatigue of these muscles during physical exercise generates many physiological reflex activation culminating in reduced blood flow to the limb muscles, resulting in decrease in muscle performance. Researchers showed that the inspiratory muscle training (IMT) is able to generate improved of athlete's physical performance. However, when it comes to wheelchair athletes there are still divergent views on the effects of IMT on the physical performance. Thus, this study aims to evaluate the effects of IMT on the physical performance and cardiorespiratory variables of wheelchair basketball players. For this purpose, the investigators will select 40 wheelchair basketball players of both genders. The participants will be allocated blindly and randomly into two groups that differ by the proposed interventions. In IMT Group, the participants will be submitted to a IMT program with inicial load of 50% of maximal inspiratory pressure (MIP); the SHAM Group will be submitted to a simulated IMT with load of 15% of MIP. All participants will pass through the same evaluation procedures before and after the interventions, so that the investagators can evaluate the benefits generated by the IMT on the physical performance and cardiorespiratory variables of wheelchair basketball players.

ELIGIBILITY:
Inclusion Criteria:

* training wheelchair basketball for more than one year.

Exclusion Criteria:

* cardiovascular or respiratory disease.
* motor or cognitive impairments that influencing the results of evaluations.
* smoking.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-01; Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Aerobic Capacity | 3 months
  The evaluation of aerobic capacity will be conducted by the 12-minutes aerobic performance test in a multisport court. In this field test the participants will have to covering the greatest distance as possible in the twelve minutes in a suitably demarcated circuit. Heart rate, blood pressure, peripheral oxygen saturation and subjective perception of effort with the Borg scale will be measured in this test.

SECONDARY OUTCOMES:
Pulmonary Function | 3 months
  The pulmonary function will be measured by a spirometer (Easy one, ndd Medizintechnik AG, Zurich, Switzerland) according to American Thoracic Society (ATS) guidelines for technique, acceptability and reproducibility.
Respiratory Muscle Strength | 3 months
  The respiratory muscle strength values will be obtained by measuring maximal inspiratory and expiratory pressures (MIP and MEP) with an analog manometer (Ger-ar®, São Paulo, Brazil) scaled in cmH2O with an operational limit of ± 300 cmH2O.
Thoracic mobility | 3 months
  The thoracic mobility will be measured by the thoracic cirtometry.
Heart rate variability | 3 months
  The heart rate variability will be measured with a Polar RS800CX® heart rate monitor (Polar Electro Co.Ltda. Kempele, Oulu, Finland).